CLINICAL TRIAL: NCT07024433
Title: Tubeless Anesthesia in Preventing Contralateral Lung Complications in Patients Undergoing Single-Port Thoracoscopic Surgery for Early-Stage Lung Cancer: A Single-Center, Prospective, Open-Label, Randomized Controlled Trial
Brief Title: Tubeless Anesthesia in Preventing Lung Complications in Patients Undergoing Surgery for Early-Stage Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024YF068-01
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer Patients
Keywords: Early-stage lung cancer; Tubeless anesthesia; Single-port thoracoscopic surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (traditional tracheal intubation group) (Other): 1. Anesthesia induction using propofol, sufentanil, and rocuronium is performed, with DLT or single-lumen tube insertion at BIS≤60 for single-lung ventilation, maintaining appropriate oxygen and ventilation parameters.
  2. Anesthesia is maintained with sevoflurane, propofol, and remifentanil, supplementing rocuronium every 30-40 minutes for muscle relaxation, with BIS maintained at 40-60.
  3. Post-surgery, ultrasound-guided thoracic paravertebral block and PCIA are used for analgesia, with extubation following standard recovery procedures.
  Interventions: Procedure: Traditional tracheal intubation
- Experimental group (Tubeless anesthesia group) (Experimental): 1. Anesthesia Induction: Implement TCI with propofol and remifentanil; insert a laryngeal mask for SIMV ventilation, and monitor vital signs including IBP and end-tidal CO2.
  2. Nerve Blocks: Perform ultrasound-guided paravertebral, pleural surface, and vagus nerve blocks using local anesthetics.
  3. Anesthesia Maintenance: Adjust remifentanil for spontaneous breathing; maintain propofol and BIS levels; manage heart rate and blood pressure with fluids and medication as needed, without using inhaled anesthetics.
  4. Postoperative Analgesia: Provide PCIA with morphine for pain management.
  Interventions: Procedure: Tubeless anesthesia

INTERVENTIONS:
Procedure: Tubeless anesthesia — 1. Anesthesia Induction: Implement TCI with propofol and remifentanil; insert a laryngeal mask for SIMV ventilation, and monitor vital signs including IBP and end-tidal CO2.
  2. Nerve Blocks: Perform ultrasound-guided paravertebral, pleural surface, and vagus nerve blocks using local anesthetics.
  3. Anesthesia Maintenance: Adjust remifentanil for spontaneous breathing; maintain propofol and BIS levels; manage heart rate and blood pressure with fluids and medication as needed, without using inhaled anesthetics.
  4. Postoperative Analgesia: Provide PCIA with morphine for pain management.
  Arms: Experimental group (Tubeless anesthesia group)
Procedure: Traditional tracheal intubation — 1. Anesthesia induction using propofol, sufentanil, and rocuronium is performed, with DLT or single-lumen tube insertion at BIS≤60 for single-lung ventilation, maintaining appropriate oxygen and ventilation parameters.
  2. Anesthesia is maintained with sevoflurane, propofol, and remifentanil, supplementing rocuronium every 30-40 minutes for muscle relaxation, with BIS maintained at 40-60.
  3. Post-surgery, ultrasound-guided thoracic paravertebral block and PCIA are used for analgesia, with extubation following standard recovery procedures.
  Arms: Control group (traditional tracheal intubation group)

SUMMARY:
The study focuses on evaluating the effectiveness and safety of tubeless anesthesia in single-port thoracoscopic surgery for early-stage lung cancer patients. Traditional anesthesia methods risk postoperative complications like lung injury and respiratory issues. Tubeless anesthesia preserves spontaneous breathing without tracheal intubation, potentially reducing these complications and enhancing recovery. The study aims to compare this technique with traditional methods, assessing its impact on contralateral lung complications, perioperative hemodynamics, complication rates, and recovery speed.

DETAILED DESCRIPTION:
With changes in lifestyle and environment, the incidence of early-stage lung cancer has been increasing annually. Traditional open surgical treatments have drawbacks such as significant trauma and noticeable pain, which has led to increased interest in minimally invasive surgery. In recent years, with continuous advancements in technology, single-port thoracoscopic surgery has become a popular choice for minimally invasive procedures, offering advantages such as minimal intraoperative trauma, mild postoperative pain, and good cosmetic results. However, traditional tracheal intubation and mechanical ventilation carry a range of potential side effects, including pressure-induced injury, lung overdistension, and the release of various pro-inflammatory mediators. Additionally, ventilator-associated lung injury occurs in about 4% of patients undergoing lung resection, with a mortality rate reaching up to 25%. The possibility of subclinical lung injury may also be underestimated. Furthermore, orotracheal and bronchial intubation can lead to various local complications, including upper respiratory tract pain, mucosal ulcers, and injury to the larynx or trachea. General anesthesia might have harmful systemic side effects, whereas local anesthesia does not pose such issues for awake patients or those with minimal sedation. Moreover, the use of muscle relaxants can lead to diaphragmatic dysfunction and atelectasis. Intravenous analgesics, especially opioids, are associated with postoperative vomiting, nausea, and respiratory depression. Importantly, postoperative pulmonary complications are among the most common complications following such surgeries, including atelectasis, lung infections, and pleural effusions, which can severely affect patient recovery and even be life-threatening. Therefore, it is crucial to find an anesthesia technique that ensures surgical efficacy while reducing postoperative pulmonary complications.

Tubeless anesthesia, which implies retaining spontaneous breathing without tracheal intubation, refers to a general anesthesia technique that does not involve tracheal intubation during thoracoscopic surgery. It employs airway devices that do not invade the trachea, alongside regional anesthesia and intravenous sedation and analgesics, to preserve spontaneous breathing. As a new anesthetic technique emerging in recent years, it offers several advantages over traditional methods, such as faster recovery, alignment with the needs of minimally invasive surgery, and a reduction in postoperative complications. Currently, the reported application range of tubeless anesthesia is extensive, encompassing simple lung biopsies, bullectomies, treatments for hyperhidrosis, as well as wedge resections, lobectomies, segmentectomies, and mediastinal tumor surgeries, even including complex tracheal tumor resections and carina reconstructions. The surgical approaches include multipoint and single-port procedures, as well as Da Vinci robotic surgeries. Although retrospective studies have confirmed the feasibility, safety, and efficacy of tubeless anesthesia in thoracoscopic-assisted minimally invasive surgery, the focus has predominantly been on the occurrence of ipsilateral lung complications.

Currently, reports on the preventive value and safety of this technique for contralateral lung complications in single-port thoracoscopic surgery in early-stage lung cancer patients are scarce, and prospective research evidence is lacking. Therefore, the primary aim of this study is to apply tubeless anesthesia in single-port thoracoscopic surgery for early-stage lung cancer patients, and to compare the incidence of contralateral lung complications three days postoperatively, perioperative hemodynamics, perioperative complication rates, and recovery speed with patients having similar baseline conditions who underwent traditional single-lumen tube + blocking tube or double-lumen tracheal intubation general anesthesia, to verify its clinical value.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤70 years;
2. ECOG performance status score 0-1;
3. Good cardiac and pulmonary function;
4. Single or multiple peripheral lung nodules planned for single-port thoracoscopic surgery, with or without mediastinal lymph node dissection or sampling;
5. Able to comply with the study visit schedule and other protocol requirements;
6. Signed informed consent and voluntary participation in the study.

Exclusion Criteria:

1. Obese patients (BMI >30);
2. Patients with difficult intubation or expected complex airway management;
3. COPD patients with copious airway secretions;
4. Patients with neurological dysfunction or who cannot cooperate while awake;
5. Patients expected to have extensive pleural adhesions or with previous lung resection;
6. Elderly and frail patients with severe hypoxia (PaO2 <60 mmHg) or hypercapnia (PaCO2 >50/55 mmHg);
7. Previous induction chemotherapy or chemoradiotherapy;
8. Intraoperative need to isolate the lung to prevent spillage and contamination of the contralateral lung;
9. Patients expected to have large surgical wounds and lengthy procedures, clinically assessed as unsuitable;
10. Patients whose cardiac and pulmonary function, or overall health, cannot withstand the procedure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Contralateral lung complications | 3 days after surgery
  This measure will determine the number of patients experiencing complications in the contralateral lung, as diagnosed through chest X-rays, within three days following surgery.

SECONDARY OUTCOMES:
Intraoperative hemodynamic analysis | During surgery
  Hemodynamic stability is monitored through three physiological parameters: heart rate (beats per minute), systolic blood pressure, and diastolic blood pressure (mmHg). During the surgery, these measurements are taken every 15 minutes, and the results for each parameter are reported in their respective units.
Intraoperative Blood Gas Analysis | The beginning and once at the end of the surgery.
  This measurement includes arterial blood gas analysis, comprising pH value, partial pressure of oxygen (PaO2 [mmHg]), partial pressure of carbon dioxide (PaCO2 [mmHg]), and bicarbonate levels (HCO3- [mmol/L]). Measurements are taken once at the beginning and once at the end of the surgery.
Consumption of Anesthetics and Vasoactive Drugs | During surgery
  The total consumption of anesthetics (measured in mg) and vasoactive drugs (measured in micrograms per kilogram per minute [mcg/kg/min]) will be documented. The data will reflect the total dosage administered during the perioperative period.
Visual Analogue Scale (VAS) for Pain Assessment | After surgery
  Pain levels will be evaluated using the Visual Analogue Scale, which ranges from 0 (no pain) to 10 (worst possible pain). Data will be collected postoperatively and presented as an average score.
Incidence of Other Adverse Reactions | Perioperative period
  Any additional adverse reactions will be recorded and categorized. The data will be presented as the number of patients experiencing specific adverse effects, along with their frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
In compliance with confidentiality requirements and to ensure the privacy of our participants, Individual Participant Data (IPD) from this clinical trial will not be shared publicly. This decision ensures adherence to ethical guidelines and legal standards for data protection, safeguarding the personal information and privacy of all participants involved in the study

REFERENCES:
- [Background] Liu Y, Liang L, Yang H. Airway management in "tubeless" spontaneous-ventilation video-assisted thoracoscopic tracheal surgery: a retrospective observational case series study. J Cardiothorac Surg. 2023 Feb 4;18(1):59. doi: 10.1186/s13019-023-02157-w. PMID 36737801
- [Background] Cui F, Liu J, Li S, Yin W, Xin X, Shao W, He J. Tubeless video-assisted thoracoscopic surgery (VATS) under non-intubated, intravenous anesthesia with spontaneous ventilation and no placement of chest tube postoperatively. J Thorac Dis. 2016 Aug;8(8):2226-32. doi: 10.21037/jtd.2016.08.02. PMID 27621880
- [Background] Kim HJ, Kim M, Park B, Park YH, Min SH. Feasibility of ventilator-assisted tubeless anesthesia for video-assisted thoracoscopic surgery. Medicine (Baltimore). 2023 Jul 14;102(28):e34220. doi: 10.1097/MD.0000000000034220. PMID 37443490
- [Background] Shao GQ, Pang DZ, Zhang JT, Wang HX, Liuru TY, Liu ZH, Liang YN, Liu JS. Spontaneous ventilation anesthesia combined with uniportal and tubeless thoracoscopic sympathectomy in selected patients with primary palmar hyperhidrosis. J Cardiothorac Surg. 2022 Jul 15;17(1):177. doi: 10.1186/s13019-022-01917-4. PMID 35840969
- [Background] Liu CY, Hsu PK, Leong KI, Ting CK, Tsou MY. Is tubeless uniportal video-assisted thoracic surgery for pulmonary wedge resection a safe procedure? Eur J Cardiothorac Surg. 2020 Aug 1;58(Suppl_1):i70-i76. doi: 10.1093/ejcts/ezaa061. PMID 32182334
- [Background] Yang LQ, Zhu L, Shi X, Miao CH, Yuan HB, Liu ZQ, Gu WD, Liu F, Hu XX, Shi DP, Duan HW, Wang CY, Weng H, Huang ZL, Li LZ, He ZZ, Li J, Hu YP, Lin L, Pan ST, Xu SH, Tang D, Sessler DI, Liu J, Irwin MG, Yu WF; POLMA-EP investigators. Postoperative pulmonary complications in older patients undergoing elective surgery with a supraglottic airway device or tracheal intubation. Anaesthesia. 2023 Aug;78(8):953-962. doi: 10.1111/anae.16030. Epub 2023 Jun 4. PMID 37270923
- [Background] Harris M, Chung F. Complications of general anesthesia. Clin Plast Surg. 2013 Oct;40(4):503-13. doi: 10.1016/j.cps.2013.07.001. Epub 2013 Aug 1. PMID 24093647
- [Background] Mullan GP, Georgalas C, Arora A, Narula A. Conservative management of a major post-intubation tracheal injury and review of current management. Eur Arch Otorhinolaryngol. 2007 Jun;264(6):685-8. doi: 10.1007/s00405-006-0234-4. Epub 2007 Mar 23. PMID 17380343
- [Background] Paudel R, Trinkle CA, Waters CM, Robinson LE, Cassity E, Sturgill JL, Broaddus R, Morris PE. Mechanical Power: A New Concept in Mechanical Ventilation. Am J Med Sci. 2021 Dec;362(6):537-545. doi: 10.1016/j.amjms.2021.09.004. Epub 2021 Sep 28. PMID 34597688
- [Background] Sakuraya M, Okano H, Masuyama T, Kimata S, Hokari S. Efficacy of non-invasive and invasive respiratory management strategies in adult patients with acute hypoxaemic respiratory failure: a systematic review and network meta-analysis. Crit Care. 2021 Nov 29;25(1):414. doi: 10.1186/s13054-021-03835-8. PMID 34844655
- [Background] Ko KJ, Lee KS. Current surgical management of pelvic organ prolapse: Strategies for the improvement of surgical outcomes. Investig Clin Urol. 2019 Nov;60(6):413-424. doi: 10.4111/icu.2019.60.6.413. Epub 2019 Oct 29. PMID 31692921
- [Background] Ichinose J, Hashimoto K, Matsuura Y, Nakao M, Okumura S, Mun M. Risk factors for bronchopleural fistula after lobectomy for lung cancer. J Thorac Dis. 2023 Jun 30;15(6):3330-3338. doi: 10.21037/jtd-22-1809. Epub 2023 Jun 5. PMID 37426169